CLINICAL TRIAL: NCT04710784
Title: The 4 Youth by Youth Project: a Pragmatic Stepped-wedge Cluster Randomized Controlled Trial to Expand Youth-friendly HIV Self-testing Services in Nigeria
Brief Title: A Pragmatic Trial to Expand Youth-friendly HIV Self-testing
Acronym: I-TEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Nigerian Institute of Medical Research (Other Government)
Responsible Party: Principal Investigator, Juliet Iwelunmor, PhD, Professor of Medicine, Washington University School of Medicine
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 31457; 4UH3HD096929 (NIH)
Record Dates: First submitted 2020-12-19; First posted 2021-01-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-07

CONDITIONS: HIV/AIDS; Sexually Transmitted Infections
Keywords: HIV Prevention; HIV Self-testing; Young people; Nigeria; 4 Youth by Youth
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- I-TEST Intervention Package (Experimental): Each study site will begin in the baseline, pre-implementation phase, and then be randomized to implement the I-TEST intervention package for a duration of three months, followed by the post-implementation phase.
  Interventions: Behavioral: Sexual health information; Behavioral: I-TEST branded HIVST package; Other: Follow-up testing and clinic assessments

INTERVENTIONS:
Behavioral: Sexual health information — We will provide participants with sexual health information, that is basic, accurate, and directly contributes to health-promoting decisions and behavior, once a week at the beginning of the study.
  Other Names: Pre-Implementation (Control Phase)
Behavioral: I-TEST branded HIVST package — The I-TEST branded HIVST package will include HIV self-testing (HIVST) kits, referral coupons, condoms, female or male hygiene products, and instructions on how to use the I-TEST photo verification App or USSD (Unstructured Supplementary Service Data) system to verify the HIVST results. Study participants will be referred to a youth-friendly health clinic for confirmatory HIV testing, STI testing (syphilis, gonorrhea, chlamydia, and hepatitis B), STI treatment and PrEP referral.
  Other Names: Intervention Implementation
Other: Follow-up testing and clinic assessments — Information to encourage routine retesting for HIV every 6 months and linkage to the youth-friendly clinic for confirmatory HIV testing, STI testing (syphilis, gonorrhea, chlamydia, and hepatitis B), STI treatment, and PrEP referral. Additionally, follow-up surveys will be administered to assess HIV testing, sexual behavior history, youth participation experience, and other related outcomes will be collected from enrolled participants.
  Other Names: Post-Implementation

SUMMARY:
The current study extends the study team's earlier efforts described in ClinicalTrail ID#: NCT04070287 and NCT03874663. The I-TEST (Innovative Tools to Expand Youth-friendly HIV Self-Testing) study known locally as the 4 Youth by Youth project, sought to develop and evaluate novel youth-friendly HIVST services in Nigeria using open challenges and apprenticeship training informed by a participatory learning collaborative model. The study thus aims to reach young Nigerians that remain undiagnosed for HIV and to facilitate linkage and retention in preventive services (includes STI testing/treatment, PrEP referral, condom use).

DETAILED DESCRIPTION:
Following the completion of the open contests and apprenticeship training, four youth teams (with four distinct interventions) were selected to undergo a one-year pilot assessment in the community. Preliminary findings from the feasibility study suggest that the youth-developed interventions have the potential to impact HIV testing as well as uptake of sexually transmitted infections (STI) testing among young people in Nigeria. As a result, the investigators identified key components from the four interventions to form a single intervention that will be evaluated in the next phase of the research. Thus, the current protocol is focused on evaluating the effectiveness of a combined, youth-developed intervention on HIV testing and other HIV prevention outcomes (i.e. condom use, PrEP referral, STI testing).

Using a stepped-wedge cluster randomized controlled trial design, the I-TEST intervention package will be implemented sequentially across 32 local government areas (LGA) whereby each LGA will be exposed to a pre-intervention (control), intervention (implementing the intervention), and post-intervention condition, according to a randomized schedule. Young people between the ages of 14-24 years will be recruited from the selected 32 local government areas through in-person events, social media platforms, and online advertisements, clinics, and community centers that cater to young people. We included two additional LGAs in November 2021 to account for civil unrest activities that are taking place across two other study sites. Due to the civil unrest, the implementation of the intervention has been affected hence the addition of the two new sites. Upon enrollment, the study team will collect baseline data on HIV testing history, sexual behavior history, youth participation experience, and other related outcomes from the study participants. Two trained youth alongside one trained supervisor will implement the I-TEST intervention at the LGAs.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-24
* Self-reported HIV negative or unknown HIV status
* Currently and planning on residing in one of the 30 areas during the next 12 months
* Able to complete the survey in English (the national language of Nigeria)
* All participants must agree to informed consent and provide their cell mobile number for follow-up and retention

Exclusion Criteria:

* Younger than 14 and older than 24
* Inability to comply with the study protocol
* Illness, cognitive impairment, or threatening behavior with acute risk to self or others
* No informed consent
* No contact phone number

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Uptake of HIV Self-testing | Up to 24 months
  The number of persons who tested with an HIV self-test. We will assess the number of persons who tested with an HIV self-test among the total number of participants in the study. The primary outcome will be ascertained using a photographic verification approach via a mobile application or a USSD (Unstructured Supplementary Service Data) system. We will also use self-reported data on HIVST results for those unable to use both systems accurately.

SECONDARY OUTCOMES:
Uptake of Facility-Based HIV testing | Up to 24 months
  The number of persons who received an HIV test at a youth-friendly clinic among the total number of participants in the study.
Sexually Transmitted Infection (STI) Testing | Up to 24 months
  The number of persons who completed a consultation at the youth-friendly clinic for STI testing. In addition, the baseline and follow-up surveys include items on knowledge and testing of sexually transmitted infections (gonorrhea, chlamydia, syphilis, and hepatitis B virus).
Sexually Transmitted Infection (STI) Treatment | Up to 24 months
  The number of persons initiating STI treatment among the total number of persons with active infection linked to care.
PrEP Referral | Up to 24 months
  PrEP referral will be assessed based on the proportion of participants who are "optimal" (assessed based on the sexual behavioral history and willingness to use PrEP) candidates for PrEP referral and the total number of participants referred for PrEP initiation at the health care facilities.
100% Condom Use | Up to 24 months
  The baseline and follow-up survey includes items on condom usage in the last sexual intercourse and a 4-item Condom Use Self Efficacy Scale.
Youth Engagement | Up to 24 months
  A 12-item scale on youth engagement will be used to assess the HIV prevention services proposed by the youth teams. The scale was adapted from the 20-item Tiffany-Eckenrode Program Participation Scale (TEPPS). Responses to the participation items were measured on a 5-point Likert-type scale, ranging from "strongly disagree (0)" to "Strongly agree (4)". Higher TEPPS scores indicate higher levels of program participation. The item is only included in the follow-up survey.
Cost effectiveness of the intervention | Up to 24 months
  The incremental cost-effectiveness ratio of participants involved in the I-TEST intervention phase compared to the control phase.

OTHER OUTCOMES:
Key Implementation Factors | Up to 24 months
  Guided by the RE-AIM framework for implementation science, semi-structured, in-depth interviews will be conducted at the individual and setting level to explore the factors associated with the implementation of the intervention (e.g., reach, adoption, implementation, and maintenance).

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Iwelunmor, PhD, Principal Investigator — St. Louis University; Oliver Ezechi, MD, Principal Investigator — Nigerian Institute of Medical Research; Joseph Tucker, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Nigerian Institute of Medical Research, Yaba, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with Saint Louis University.
Supporting Information: SAP

REFERENCES:
- [Background] WHO/TDR. (2018). Crowdsourcing in Health and Health Research: A Practical Guide (TDR/STRA/18.4). Retrieved from Geneva: https://www.who.int/tdr/publications/year/2018/crowdsourcing-practical-guide/en/
- [Background] Iwelunmor J, Ezechi O, Obiezu-Umeh C, Gbaja-Biamila T, Nwaozuru U, Oladele D, Musa AZ, Idigbe I, Uzoaru F, Airhihenbuwa C, Muessig K, Conserve DF, Kapogiannis B, Tucker JD. The 4 youth by youth HIV self-testing crowdsourcing contest: A qualitative evaluation. PLoS One. 2020 May 29;15(5):e0233698. doi: 10.1371/journal.pone.0233698. eCollection 2020. PMID 32469971
- [Background] Saunders AN. Incubator noise: a method to decrease decibels. Pediatr Nurs. 1995 May-Jun;21(3):265-8. PMID 7792110
- [Background] Cincotta FA. Dental anesthesia: the private office versus the hospital. Dent Surv. 1980 Aug;56(8):20-1. No abstract available. PMID 6935128
- [Derived] Iwelunmor J, Obiezu-Umeh C, Gbaja-Biamila T, Oladele D, Nwaozuru U, Musa AZ, Abodunrin OR, Akinsolu FT, Ojo T, Olusanya O, Bamidele T, Ezeama N, Okeke C, Johnny I, Ekene M, Rahman N, Musari-Martins T, Ajibaye S, Lateef A, Ojo V, Babatunde Y, Airhihenbuwa CO, Muessig K, Rosenberg N, BeLue R, Xian H, Conserve DF, Zou Z, Ong JJ, Zhang L, Curley J, Nkengasong S, Mason S, Tang W, Bayus B, Ogedegbe G, Tucker JD, Ezechi O. The 4 youth by youth (4YBY) crowdsourced HIV prevention intervention: A stepped-wedge longitudinal trial on HIV self-testing uptake among adolescents and young people in Nigeria. Contemp Clin Trials. 2025 Jul;154:107919. doi: 10.1016/j.cct.2025.107919. Epub 2025 Apr 20. PMID 40262659
- [Derived] Anikamadu O, Ezechi O, Engelhart A, Nwaozuru U, Obiezu-Umeh C, Ogunjemite P, Bale BI, Nwachukwu D, Gbaja-Biamila T, Oladele D, Musa AZ, Mason S, Ojo T, Tucker J, Iwelunmor J. Expanding Youth-Friendly HIV Self-Testing Services During the COVID-19 Pandemic: Qualitative Analysis of a Crowdsourcing Open Call in Nigeria. JMIR Form Res. 2024 Apr 30;8:e46945. doi: 10.2196/46945. PMID 38687582
- [Derived] Iwelunmor J, Tucker JD, Obiezu-Umeh C, Gbaja-Biamila T, Oladele D, Nwaozuru U, Musa AZ, Airhihenbuwa CO, Muessig K, Rosenberg N, BeLue R, Xian H, Conserve DF, Ong JJ, Zhang L, Curley J, Nkengasong S, Mason S, Tang W, Bayus B, Ogedegbe G, Ezechi O. The 4 Youth by Youth (4YBY) pragmatic trial to enhance HIV self-testing uptake and sustainability: Study protocol in Nigeria. Contemp Clin Trials. 2022 Mar;114:106628. doi: 10.1016/j.cct.2021.106628. Epub 2021 Nov 17. PMID 34800699
- See also: 4 Youth by Youth Website — https://4yby.org/
- See also: SESH Crowdsourcing Clinic — https://www.seshglobal.org/